CLINICAL TRIAL: NCT06592001
Title: Assessment of a Chronically Implanted Parasternally Delivered EV-ICD Lead (ASCEND EV) Study
Acronym: ASCEND EV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AtaCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOC-10280
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Ventricular Arrythmia; Ventricular Fibrillation; Ventricular Tachycardia
Keywords: Ventricular Defibrillation; Extravascular
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AtaCor EV-ICD Lead System (Experimental): Subjects implanted with the Atala™ lead
  Interventions: Device: Atala™ lead

INTERVENTIONS:
Device: Atala™ lead — Subjects will receive the Atala™ lead being evaluated in the study.
  Other Names: AtaCor EV-ICD Atala™ lead; AtaCor Atala™ lead

SUMMARY:
The ASCEND EV Study is a prospective, multi-center, single-arm, non-randomized study without concurrent or historical controls. The purpose of the study is to evaluate the Investigational Devices through at least 3-months of follow-up to inform the design of a subsequent pivotal clinical investigation.

The objectives of the study are to: 1) preliminarily validate safety and effectiveness of the Atala™ lead as a permanent ICD lead when used with a compatible ICD pulse generator, 2) evaluate suitability of clinical study testing methods and 3) inform statistically powered primary safety and effectiveness endpoints in a subsequent pivotal clinical investigation.

DETAILED DESCRIPTION:
The primary safety endpoint is freedom from major Adverse Device Effects (ADEs) through 3-months. The primary performance endpoint is successful induced ventricular arrhythmia (IVA) test in the final system configuration.

Up to three (3) Investigational Sites will participate with up to 35 Subjects enrolled in the study. Subjects who meet current indications for ICD therapy will be eligible for participation. Eligible Subjects will receive an Atala™ lead connected to a commercially available ICD positioned in a left pectoral or left lateral location.

The Atala™ lead will be connected to a compatible ICD pulse generator and tested to verify appropriate sensing and defibrillation. Abbreviated IVA testing will be performed at the 3-month follow-up visit to verify continued sensing and defibrillation effectiveness. Starting at 6 months, Subjects will be followed every 6 months until the study is closed. The study is expected to remain open for at least 3 years.

Endpoints will be analyzed and summarized in a final study report after all active Subjects have completed the 3-month visit.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Class I or IIa indication for implantation of an ICD according to the ACC/AHA/HRS Guidelines or ESC guidelines

Exclusion Criteria:

1. Participation in any concurrent clinical study without prior written approval from the Sponsor
2. Inability or unwillingness to provide informed consent to participate in the Study
3. Any known conditions which may complicate the AtaCor EV-ICD Lead System implant procedure or prevent the subject from completing protocol testing through the 3-month follow-up visit
4. Circumstances that may prevent data collection or completion of specified follow-up visits
5. Allergies to any device materials listed in the Instructions for Use (IFU)
6. Subjects on anticoagulation therapy that cannot be temporarily discontinued for the procedure
7. Known history of lung disease with FEV1 < 1.0 Liter

   Device Related:
8. Presence or planned use of medical devices that introduce current into the body (e.g., pacemaker, LVAD, neurostimulator, etc.)
9. Implanted with or planned implantation of any device which delivers current in the body, that may interfere with therapy delivery, including, but not limited to a pacemaker, or neurostimulator
10. Presence or planned use of a subcutaneous ICD lead, subcutaneous coils/arrays, epicardial patches or epicardial pace/sense leads
11. Any known need for future MRI

    Anatomy Related:
12. BMI ≥ 35 kg/m2
13. Structural abnormalities of the heart that may increase risk of the study procedure or an obstructed/restricted pathway into the mediastinum
14. Prior sternotomy of any type, including but not limited to median, mini or clamshell
15. Prior surgery with disruption of the lung, pericardium or connective tissue between the sternum and pericardium
16. Known significant anatomic derangement of or within the thorax (e.g., pectus excavatum, significant scoliosis) and associated with displacement of the heart or lungs or impeded mediastinal access.
17. History of thoracic radiation therapy, pneumothorax, pneumomediastinum or other medical treatments/conditions which may complicate the AtaCor EV-ICD Lead System implant procedure
18. Known adhesions in the thorax or history of medical treatments, surgeries or conditions that increase the potential for adhesions in the thorax
19. Surgically corrected congenital heart disease (not including catheter-based procedures)

    Cardiac Related:
20. Subjects who require permanent bradycardia pacing or cardiac resynchronization therapy
21. NYHA IV functional class in past 90 days
22. Inotropic therapy in past 180 days
23. Known history of pericardial disease, pericarditis or mediastinitis
24. Patients with a medical condition that precludes them from undergoing defibrillation testing:

    * Severe aortic stenosis
    * Current Intracardiac LA or LV thrombus
    * Severe proximal three-vessel or left main coronary artery disease without revascularization
    * Hemodynamic instability
    * Unstable angina
    * Recent stroke or transient ischemic attack (within the last 6 months)
    * Known inadequate external defibrillation
    * LVEF < 20%
    * LVEDD >70 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from major ADEs | Through 3 months post-implant
  Freedom from major Adverse Device Effects (ADEs)
Successful IVA Test | At the time of procedure
  Successful induced ventricular arrhythmia (IVA) test in the final system configuration

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospital Center Split, Split, Croatia
- Christchurch Hospital, Christchurch, New Zealand
- Sanatorio Italiano, Asunción, Paraguay